CLINICAL TRIAL: NCT00479583
Title: A Phase I Study to Determine the Safety, Pharmacokinetics and Pharmacodynamics of BMS-690514 in Combination With FOLFIRI and FOLFOX in Subjects With Advanced Metastatic Solid Tumors
Brief Title: Combination Trial of BMS-690514 in Combination With FOLFIRI and FOLFOX
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA187-005
Record Dates: First submitted 2007-05-24; First posted 2007-05-28 (Estimated); Last update posted 2011-11-30 (Estimated); Status verified 2011-03

CONDITIONS: Cancer
Keywords: Cancer (solid tumors)
MeSH Terms: conditions — Neoplasms | interventions — BMS-690514; Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: BMS-690514 / FOLFIRI
- B (Active Comparator)
  Interventions: Drug: BMS-690514 / FOLFOX

INTERVENTIONS:
Drug: BMS-690514 / FOLFIRI — Tablets / IV, Oral / IV, up to 200 mg / irinotecan 180mg/m2, leucovorin 400 mg/m2, 5FU 400mg/m2 bolus, 2400 mg/m2 inf, once daily / q 2 weeks, up to 24 mos
  Arms: A
Drug: BMS-690514 / FOLFOX — Tablets / IV, Oral / IV, up to 200 mg / oxaliplatin 85 mg/m2, leucovorin 400 mg/m2, 5FU 400mg/m2 bolus, 2400 mg/m2 inf, once daily / q 2 weeks, up to 24 mos
  Arms: B

SUMMARY:
The purpose of this research study is to determine the highest dose of BMS-690514 that can be safely given in combination with the chemotherapeutic regimens (FOLFIRI and FOLFOX) to patients with advanced cancer

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for FOLFIRI or FOLFOX therapy
* ECOG performance status score 0-1
* At least 4 weeks since the last chemotherapy, immunotherapy or radiotherapy with:
* At least 4 weeks since anti-cancer hormonal therapy OR targeted therapy (for instance tamoxifen or Tarceva)
* No maximum age for Study Arm A (FOLFOX)
* 18-65 years of age for Study Arm B (FOLFIRI)

Exclusion Criteria:

* Treatment with other TKIs within the past 4 weeks
* Active inflammatory bowel disease
* Major gastrointestinal surgery which may affect absorption of the drug, any surgery within the last 4 weeks
* History of thromboembolism
* Severe unmanageable diarrhea
* Uncontrolled or significant cardiovascular disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-09; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Safety assessment | throughout the study
dose-limiting toxicity (DLT) | assessed for individual patients from C1D1 to C1D28 during the dose escalation portion of the protocol, until maximum tolerated dose is identified
determination of maximum tolerated dose (MTD) | during dose escalation portion of the protocol. Three to six subjects are treated at a specified dose level. If deemed safe dose escalation continues until the maximum tolerated dose is identified

SECONDARY OUTCOMES:
Describe anti-tumor of combination therapy | Every 8 weeks throughout the study
Describe effects of combination therapy on markers of therapeutic activity. e.g. blood, plasma and biopsy samples | throughtout the study

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (4):
- United States (2):
  - University Of Alabama At Birmingham, Birmingham, Alabama
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
- France (2):
  - Local Institution, Saint-Herblain
  - Local Institution, Villejuif

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx